CLINICAL TRIAL: NCT03398837
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase 3 Trial to Evaluate Efficacy and Safety of Lenabasum in Diffuse Cutaneous Systemic Sclerosis
Brief Title: Trial to Evaluate Efficacy and Safety of Lenabasum in Diffuse Cutaneous Systemic Sclerosis
Acronym: RESOLVE-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor terminated open-label extension
Sponsor: Corbus Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JBT101-SSc-002
Record Dates: First submitted 2018-01-05; First posted 2018-01-16 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Diffuse Cutaneous Systemic Sclerosis
Keywords: Scleroderma; cannabinoid receptor type 2 agonist; anabasum; JBT-101; lenabasum
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — lenabasum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Lenabasum 5 mg BID
  Interventions: Drug: Lenabasum 5 mg
- Cohort 2 (Experimental): Lenabasum 20 mg BID
  Interventions: Drug: Lenabasum 20 mg
- Cohort 3 (Placebo Comparator): Placebo BID
  Interventions: Other: Placebo oral capsule

INTERVENTIONS:
Drug: Lenabasum 5 mg — Subjects will receive lenabasum 5 mg twice daily.
  Arms: Cohort 1
Drug: Lenabasum 20 mg — Subjects will receive lenabasum 20 mg twice daily.
  Arms: Cohort 2
Other: Placebo oral capsule — Subjects will receive placebo twice daily.
  Arms: Cohort 3

SUMMARY:
This is a Phase 3 multicenter, double-blind, randomized, placebo-controlled study assessing the efficacy and safety of lenabasum for the treatment of diffuse cutaneous systemic sclerosis (SSc). Approximately 354 subjects will be enrolled in this study at about 60 sites in North America, Europe, Australia, and Asia. The planned duration of treatment with study drug is 52 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

1. ≥ 18 years of age at the time Informed Consent is signed.
2. Diffuse cutaneous SSc (skin thickening on upper arms, upper legs, or trunk).
3. Disease duration ≤ 6 years from the first non-Raynaud's symptom.
4. No new or increased doses of immunosuppressive medications within 8 weeks prior to Screening.

Key Exclusion Criteria:

1. Unstable SSc or SSc with end-stage organ involvement at Screening or Visit 1.
2. Any of the following values for laboratory tests at Screening:

   1. A positive pregnancy test in women of childbearing potential;
   2. Hemoglobin < 9 g/dL for males and < 8 g/dL for females;
   3. Neutrophils < 1.0 ×10^9/L;
   4. Platelets < 75 ×10^9/L;
   5. Creatinine clearance < 50 mL/min according to the Modification of Diet in Renal Disease (MDRD) Study equation;
   6. Aspartate aminotransferase or alanine aminotransferase > 2.0 × upper limit of normal.
3. Any medical condition or concurrent medical therapies at Screening or Visit 1, including a history of non-compliance with medical treatments, that may put the subject at greater safety risk, influence response to study product, or interfere with study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Efficacy of lenabasum compared to placebo for the American College of Rheumatology Combined Response Index in diffuse cutaneous Systemic Sclerosis score. | American College of Rheumatology Combined Response Index score through study completion, up to 1 year.
  The ACR CRISS exponential algorithm determines the predicted probability of improvement from baseline, incorporating change in mRSS, FVC % predicted, physician and patient global assessments, and HAQ-DI. The outcome is a continuous variable between 0.0 and 1.0 (0 - 100%). A higher score indicates greater improvement.

SECONDARY OUTCOMES:
Efficacy of lenabasum compared to placebo for the change from baseline in modified Rodnan skin score. | Change from baseline through study completion, up to 1 year.
  mRSS evaluates a subject's skin thickness on a 4 point scale for 17 surface anatomic areas: 0 = normal skin; 1 = mild thickness; 2 = moderate thickness; 3 = severe thickness with inability to pinch skin into fold. The individual values of the 17 surface areas are summed to define the total skin score with a maximum score of 51.
Efficacy of lenabasum compared to placebo for the change from baseline in Health Assessment Questionnaire - Disability Index. | Change from baseline through study completion, up to 1 year.
  It includes 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities. There are 2 or 3 questions for each section. Scoring within each section is from 0 (without any difficulty) to 3 (unable to do). The individual scores of the eight sections are summed and divided by 8. The result is the disability index or functional disability index. A higher score indicates more functional disability.
Efficacy of lenabasum compared to placebo for the change from baseline in forced vital capacity. | Change from baseline through study completion, up to 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Spiera, MD, Principal Investigator — Professor of Clinical Medicine, Weill Cornell Medical College; Chris Denton, MD, Principal Investigator — Professor of Experimental Rheumatology and Consultant Rheumatologist and Centre Head, Royal Free Hospital
Locations (74):
- United States (27):
  - University of California San Diego, La Jolla, California
  - Pacific Arthritis Care Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - Tulane University Medical Center, New Orleans, Louisiana
  - John Hopkins University, Scleroderma Center, Baltimore, Maryland
  - Massachusetts General Hospital, Division of Rheumatology, Boston, Massachusetts
  - Boston University Medical Center (BUMC) - General Clinical Research Unit (GCRU), Boston, Massachusetts
  - Michigan Medicine, Ann Arbor, Michigan
  - University of Minnesota Health Clinical Research Unit, Minneapolis, Minnesota
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Rutgers Clinical Research Center, Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - The Steffens Scleroderma at The Center for Rheumatology, Albany, New York
  - Columbia University Medical Center, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Toledo, Toledo, Ohio
  - University of Pennsylvania Health System - PCAM, Dept. of Rheumatology, Philadelphia, Pennsylvania
  - UPMC Arthritis and Autoimmunity Center, Falk Clinic, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Metroplex Clinical Research Center, Dallas, Texas
  - UTP Rheumatology Clinic, Houston, Texas
  - University of Utah Hospitals and Clinics, Salt Lake City, Utah
  - Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin
- Australia (4):
  - Royal Adelaide Hospital, Adelaide
  - Liverpool Hospital, Liverpool
  - St Vincent's Hospital, Melbourne
  - Royal Prince Alfred Hospital, Sydney
- Canada (2):
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal
  - The Arthritis Centre, Winnipeg
- Germany (8):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Charité- Universitätsmedizin Berlin, Klinik für Rheumatologie und Klinische Immunologie, Abteilung -Neue Therapien & Studien-, Berlin
  - University Hospital Cologne, Department of Dermatology and Venereology, Cologne
  - Universitätsklinik Köln,Klinik und Poliklinik für Dermatologie und Venerologie, Cologne
  - Department of Internal Medicine 3, University of Erlangen-Nuremberg, Erlangen
  - University Medical Center Freiburg, Freiburg im Breisgau
  - Kerckhoff-Klinik GmbH, Zentrum Rheumatologie u. Klin. Immunologie, Studienambulanz, Nauheim
  - University Hospital Ulm, Ulm
- Israel (4):
  - Rambam Health Corporation, Haifa
  - Bnai Zion Medical Center, Haifa
  - Meir Medical Center - Internal Medicine E, Kfar Saba
  - Sheba Medical Center, Ramat Gan
- Japan (8):
  - Kyushu University Hospital, Fukuoka
  - Kanazawa University Hospital, Kanazawa
  - Gunma University Hospital, Maebashi
  - Hokkaido University Hospital, Sapporo
  - National University Corporation Tohoku University Tohoku University Hospital, Sendai
  - Osaka University Hospital, Suita
  - Nippon Medical School Hospital, Tokyo
  - Yokohama City University Hospital, Yokohama
- Netherlands (3):
  - Leiden University Medical Center, Leiden, South Holland
  - Erasmus Medical Center, Rotterdam
  - Haga Hospital, The Hague
- Poland (3):
  - Samodzielny Publiczny Szpital Kliniczny nr 1; Katedra i Klinika Dermatologii, Wenerologii i Dermatologii Dziecięcej Uniwersytetu Medycznego w Lublinie, Lublin
  - Medyczne Centrum Hetmanska, Poznan
  - Reum-Medica S.C, Wroclaw
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Hanyang University Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (2):
  - Hospital Universitari de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Doctor Peset, Valencia
- Switzerland (2):
  - Cantonal Hospital St. Gallen, Sankt Gallen
  - University Hospital Zurich, Zurich
- United Kingdom (7):
  - Ninewells Hospital, Dundee, Scotland
  - Freeman Hospital, Newcastle, Tyne and Wear
  - Russell's Hall Hospital, Dudley, West Midlands
  - Leeds Institute of Rheumatic and Musculoskeletal Medicine (LIRMM), Leeds
  - Royal Free Hospital London NHS Foundation Trust, London
  - Guy's and St.Thomas' NHS Foundation Trust, London
  - Salford Royal NHS Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: Undecided